CLINICAL TRIAL: NCT03250234
Title: Influence of Carbohydrate Availability on Skeletal Muscle and Circulating microRNA Expression
Brief Title: Carbohydrate Availability and microRNA Expression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17-17H
Record Dates: First submitted 2017-07-19; First posted 2017-08-15 (Actual); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Glycogen Depletion
Keywords: microRNA, carbohydrate oxidation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adequate Carbohydrate (Other): Carbohydrate beverage (1 g/kg/hr) Adequate carbohydrate diet 6.0 g/kg/d
  Interventions: Other: Adequate Carbohydrate
- Low Carbohydrate (Other): Non-nutritive control beverage. Low carbohydrate diet 1.2 g/kg/d
  Interventions: Other: Low Carbohydrate

INTERVENTIONS:
Other: Adequate Carbohydrate — During the 3-hr recovery period after glycogen depletion participants will consume a carbohydrate (1 g/kg/hr) beverage For the day participants will consume a diet of 6.0 g/kg/d carbohydrate following glycogen depletion
  Arms: Adequate Carbohydrate
Other: Low Carbohydrate — During the 3-hr recovery period after glycogen depletion participants will consume a nutrient free beverage.
  For the day participants will consume a diet of 1.2 g/kg/d carbohydrate following glycogen depletion
  Arms: Low Carbohydrate

SUMMARY:
This investigation will examine the impact of skeletal muscle glycogen stores on skeletal muscle and circulating microRNA expression and exogenous carbohydrate oxidation.

Primary Objective Determine the influence of carbohydrate availability (e.g., glycogen depletion and repletion) on skeletal muscle microRNA expression, and if changes in circulating microRNA are reflective of changes in skeletal muscle microRNA.

Secondary Objective Determine how initiation of exercise with adequate or low glycogen stores effects exogenous carbohydrate efficiency.

DETAILED DESCRIPTION:
Twelve, normal weight, healthy, physically active men and women will complete a glycogen depletion protocol, cycling at various intensities until failure. Participants will then consume a carbohydrate (CHO: 1 g/kg/hr) or an energy free control (CON) beverage matched for taste and color during the first 3-hr post glycogen depletion. For the remainder of the day participants will consume a diet designed to adequately (6.0 g CHO/kg/d) or inadequately (1.2 g CHO/kg/d) replenish glycogen stores. The following day participants will to complete 80-min of steady-state (~60% VO2peak) cycle ergometry consuming carbohydrate at a rate of 1.8 g/min enriched with a stable isotope of carbon to determine exogenous carbohydrate efficiency when glycogen stores are low or adequate at the onset of exercise.

Following a minimum 7-d washout period volunteers will return to the laboratory to complete the second arm of the investigation. To ensure glycogen stores are similar between volunteers on testing day, 48-hrs prior to testing all volunteers will complete a glycogen depletion protocol and then consume a diet providing 6.0 g/kg/d carbohydrate to replenish glycogen stores.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 39 years
* Weight stable (±5 lbs) for at least 2 months prior to the start of the study
* Body mass index (BMI) between 18.5-30 kg/m2
* Recreationally active based on assessment of physical activity history 2-4 days per week aerobic and/or resistance exercise
* Refrain from taking any NSAIDS (i.e., aspirin, Advil®, Aleve®, Naprosyn®, or any aspirin-containing product for 10 days before and at least 5 days AFTER each muscle biopsy. (*Tylenol® or acetaminophen is ok to use if needed for discomfort)
* Refrain from the use of alcohol and nicotine for the duration of the study
* Females must be on contraception (e.g., oral birth control, NuvaRing®, Depo Provera®, etc.)
* Supervisor approved leave status for federal civilian employees working within the US Army Natick Soldier Systems Center

Exclusion Criteria:

* Metabolic or cardiovascular abnormalities, gastrointestinal disorders (i.e., kidney disease, diabetes, cardiovascular disease, etc.)
* Disease or medication (i.e., diabetes medications, statins, corticosteroids, etc) that affects macronutrient utilization and/or the ability to participate in strenuous exercise
* Allergies or intolerance to foods (including but not limited to lactose intolerance/milk allergy), vegetarian practices, or medications (including, but not limited to, lidocaine or phenylalanine) to be utilized in the study
* Anemia (HCT < 38) and Sickle Cell Anemia/Trait
* Abnormal prothrombin time (PT)/ partial thromboplastin time (PTT) test or problems with blood clotting
* Present condition of alcoholism, use of nutritional/sports supplements, anabolic steroids, or other substance abuse issues
* Musculoskeletal injuries that compromise the ability to exercise
* Blood donation within 8 weeks of beginning the study
* Pregnancy

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- USARIEM, Natick, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a cross over design. 12 participants enrolled and completed both study arms.
Groups:
- Adequate Carbohydrate First, Then Low Carbohydrate: Carbohydrate beverage (1 g/kg/hr) Adequate carbohydrate diet 6.0 g/kg/d first, then Low carbohydrate diet 1.5 g/kg/d
  Adequate Carbohydrate: During the 3-hr recovery period after glycogen depletion participants will consume a carbohydrate (1 g/kg/hr) beverage For the day participants will consume a diet of 6.0 g/kg/d carbohydrate following glycogen depletion
  7 day washout
  Low Carbohydrate: During the 3-hr recovery period after glycogen depletion participants will consume a nutrient free (0 kcal) beverage For the day participants will consume a diet of 1.5 g/kg/d carbohydrate following glycogen depletion
- Low Carbohydrate First, Then Adequate Carbohydrate: Non-nutritive control beverage. Low carbohydrate diet 1.5 g/kg/d first, then adequate carbohydrate diet 6.0 g/kg/d
  Low Carbohydrate: During the 3-hr recovery period after glycogen depletion participants will consume a nutrient free (0 kcal) beverage.
  For the day participants will consume a diet of 1.5 g/kg/d carbohydrate following glycogen depletion
  7 day washout
  Adequate Carbohydrate: During the 3-hr recovery period after glycogen depletion participants will consume a carbohydrate (1 g/kg/hr) beverage For the day participants will consume a diet of 6.0 g/kg/d carbohydrate following glycogen depletion
Period: Overall Study
Arm/Group | Adequate Carbohydrate First, Then Low Carbohydrate | Low Carbohydrate First, Then Adequate Carbohydrate
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Adequate Carbohydrate First, Then Low Carbohydrate: Carbohydrate beverage (1 g/kg/hr) Adequate carbohydrate diet 6.0 g/kg/d
  Adequate Carbohydrate: During the 3-hr recovery period after glycogen depletion participants will consume a carbohydrate (1 g/kg/hr) beverage For the day participants will consume a diet of 6.0 g/kg/d carbohydrate following glycogen depletion
- Low Carbohydrate First, Then Adequate Carbohydrate: Non-nutritive control beverage. Low carbohydrate diet 1.5 g/kg/d
  Low Carbohydrate: During the 3-hr recovery period after glycogen depletion participants will consume a nutrient free beverage.
  For the day participants will consume a diet of 1.5 g/kg/d carbohydrate following glycogen depletion
- Total: Total of all reporting groups
Arm/Group | Adequate Carbohydrate First, Then Low Carbohydrate | Low Carbohydrate First, Then Adequate Carbohydrate | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: This was a crossover study
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 6 | 6 | 12
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This was a crossover study
  Participants
    Female | 0 | 0 | 0
    Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Population: This was a crossover study
  Participants
    United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Fold Change in microRNA Expression From Baseline
Description: Determine the influence of low or adequate glycogen on expression of skeletal muscle and circulating microRNA. Expression of microRNA was determined using real time polymerase chain reaction analysis. microRNA expressions were calculated as a fold change relative to baseline.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: fold change
Groups:
- Low Carbohydrate: Non-nutritive control beverage. Low carbohydrate diet 1.5 g/kg/d
  Low Carbohydrate: During the 3-hr recovery period after glycogen depletion participants will consume a nutrient free (0 kcal) beverage.
  For the day participants will consume a diet of 1.5 g/kg/d carbohydrate following glycogen depletion
Arm/Group | Adequate Carbohydrate | Low Carbohydrate
Number analyzed (Participants) | 12 | 12
fold change | 0.73 (.2) | 1.36 (1.35)

2. Secondary Outcome: Exogenous Carbohydrate Oxidation
Description: Determine how initiation of exercise with adequate or low glycogen stores effects exogenous carbohydrate efficiency. Exogenous carbohydrate oxidation was measured using an oral 13C-glucose isotope that was consumed in the study carbohydrate drink during steady-state cycling. Breath samples were collected during exercise and analyzed using isotope ratio mass spectrometry to calculate exogenous carbohydrate oxidation rates.
Time Frame: 80 minutes
Measure: Mean (Standard Deviation); unit: g/min
Arm/Group | Adequate Carbohydrate | Low Carbohydrate
Number analyzed (Participants) | 12 | 12
g/min | .87 (.16) | .84 (.14)

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Hamstring cramping
Arm/Group | Adequate Carbohydrate | Low Carbohydrate
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adequate Carbohydrate (N=12) | Low Carbohydrate (N=12)
Hamstring Cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT03250234/Prot_SAP_000.pdf